CLINICAL TRIAL: NCT06763718
Title: Optimizing Fitness: Post Bariatric Surgery With Modified Qigong Breathing Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Collaborators: Al-Zaytoonah University of Jordan (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Ahmed Abd El hady El Fahl,ph.d, Assi.Prof.Dr.Ahmed Mohamed Ahmed Abd elhady Elfahl, Al-Zaytoonah University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005533
Record Dates: First submitted 2024-12-31; First posted 2025-01-08 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Bariatric Surgery
Keywords: Fitness; Bariatric Surgery; Qigong Breathing Exercise

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Sham Comparator): No exercise will be given to the participants in the control group
  Interventions: Other: Control
- Modified Qigong Breathing Exercise (Experimental): The exercise is recommended to be performed standing, or modified standing with trunk leaning forward and bilateral upper extremities support on countertop. Initial position: Stand up with feet shoulder-width apart, hands down along your body, or put palms on the abdomen. Take a deep breath, squaring shoulders, and pull in belly at the same time. Hold breath for 3 to 4 seconds, while keeping abdomen retracted with maximally contracting abdominal muscles. Exhale, so the shoulders go back to the starting position, while chest and abdominal muscles relax. Repeat this exercise 10 times. Note. If the stomach is difficult to draw in a standing position, it is possible to perform the exercise with both hands resting on support.
  Interventions: Other: Modified Qigong Breathing Exercise

INTERVENTIONS:
Other: Modified Qigong Breathing Exercise — The exercise is recommended to be performed standing, or modified standing with trunk leaning forward and bilateral upper extremities support on countertop. Initial position: Stand up with feet shoulder-width apart, hands down along the body, or put palms on the abdomen. Take a deep breath, squaring shoulders, and pull in belly at the same time. Hold breath for 3 to 4 seconds, while keeping abdomen retracted with maximally contracting abdominal muscles. Exhale, so the shoulders go back to the starting position, while chest and abdominal muscles relax. Repeat this exercise 10 times. Note. If the stomach is difficult to draw in a standing position, it is possible to perform the exercise with both hands resting on support.
  Duration: 30 minutes, 3 days/ week for 8 weeks
  Arms: Modified Qigong Breathing Exercise
Other: Control — No exercise will be given to the participants in the control group
  Arms: Control

SUMMARY:
Bariatric surgery has been reported to be the most effective treatment option for losing and maintaining body weight and improving comorbidities and mortality associated with morbid obesity. Nevertheless, even though physical activity is recommended to optimize bariatric surgery results. Very little is known, about whether engaging in an exercise program after surgery can provide additional improvement in health outcomes. While to date there are relatively few researches studied the effect of exercise in patients who have undergone bariatric surgery. This study was conducted to explore the influence of Modified Qigong Breathing Exercise on pulmonary function, endurance and fitness on post bariatric surgery patients.

Qigong as ancient Chinese traditional medicine have been documented to be effective in treating obesity. Literature showing that the desire to eat and the feeling of hunger, along with prospective food consumption in patients with obesity.

DETAILED DESCRIPTION:
Bariatric surgery has been reported to be the most effective treatment option for losing and maintaining body weight and improving comorbidities and mortality associated with morbid obesity. Nevertheless, even though physical activity is recommended to optimize bariatric surgery results. Very little is known, about whether engaging in an exercise program after surgery can provide additional improvement in health outcomes. While to date there are relatively few researches studied the effect of exercise in patients who have undergone bariatric surgery. This study was conducted to explore the influence of Modified Qigong Breathing Exercise on pulmonary function,endurance and fitness on post bariatric surgery patients.

Bariatric surgery has been reported to be the most effective treatment option for losing and maintaining body weight and improving comorbidities and mortality associated with morbid obesity. Nevertheless, even though physical activity is recommended to optimize bariatric surgery results. Very little is known, about whether engaging in an exercise program after surgery can provide additional improvement in health outcomes. While to date there are relatively few researches studied the effect of exercise in patients who have undergone bariatric surgery.

Qigong as ancient Chinese traditional medicine have been documented to be effective in treating obesity. Literature showing that the desire to eat and the feeling of hunger, along with prospective food consumption in patients with obesity .

ELIGIBILITY:
Inclusion Criteria:

* Both male and fem
* age ranged from 18-25 years old
* at least 6 months after BS

Exclusion Criteria:

* Patients with nerve root compression
* spine disorders
* spinal fracture
* previous spinal surgery
* pregnancy
* lower limb injury
* Any contraindication to the exercise therapy

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2025-01-05 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Pulmonary function by (SP - electronic hand held spirometer) | at base line and 8 weeks
  Forced vital capacity (FVC) [Time Frame: 8 weeks]
Core endurance by McGill tests | At base line and 8 weeks
  trunk anterior flexor test
Pulmonary function by (SP - electronic hand held spirometer) | at base line and 8 weeks
  forced expiratory volume in 1 second (FEV1) [Time Frame: 8 weeks]
Pulmonary function by (SP - electronic hand held spirometer) | at base line and 8 weeks
  Peak expiratory flow (PEF) [Time Frame: 8 weeks]
Core endurance by McGill tests | at base line and 8 weeks
  trunk posterior extensor test
Core endurance by McGill tests | at base line and 8 weeks
  the right lateral plank

SECONDARY OUTCOMES:
Resting metabolic rate | at base line and 8 weeks
  Change in resting metabolic rate measured by indirect calorimetry at 0 and 8 weeks.
Percent fat mass | at base line and 8 weeks
  Change in fat mass percentage measured by DXA at 0 and 8 weeks
Weight measurement | ate base line and 8 weeks
  Weight measurement in kilogram
Height measurement | at base line and 8 weeks
  Height measurement in centimeter

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of ohysical therapy Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
not be shared

REFERENCES:
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC4888907/